CLINICAL TRIAL: NCT03525704
Title: Evaluation of Contact Lens Saline Solutions With Scleral GP Contact Lens Wearers Experiencing Fogging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contamac Ltd (Industry)
Collaborators: Andre Vision and Device Research (Unknown); The Contact Lens Center at Optique (Unknown); Premiere Vision Group (Unknown); Havasu Eye Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AVDR 2018-01 v1.2
Record Dates: First submitted 2018-03-30; First posted 2018-05-16 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Contact Lens Complication; Debris in Post Lens Tear Reservoir
Keywords: Fogging; Insertion Solutions; RGP; Scleral; Contact Lenses

STUDY DESIGN:
Intervention Model Description: One-month, approximately 36 subjects enrolled (~12/site), randomized, double-masked crossover trial.
Who Masked: Participant, Investigator
Masking Description: Randomized, Double-Masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Saline Solution Enriched (Experimental): Saline Solution enriched with electrolytes and PH balanced to mimic normal tears
  Interventions: Device: Saline Solution Enriched
- Saline Rinse Solution (Active Comparator): Saline Solution .9% NaCL
  Interventions: Device: Saline Rinse Solution

INTERVENTIONS:
Device: Saline Solution Enriched — Sterile single dose, Preservative Free, PH Balanced, Enriched with IONs rinsing and Insertion Solution
  Other Names: NutriFill; GatorFill
  Arms: Saline Solution Enriched
Device: Saline Rinse Solution — sterile unit dose non-preserved, 0.9% NaCl (normal saline) solution i
  Other Names: LacriPure; ScleralFil
  Arms: Saline Rinse Solution

SUMMARY:
Evaluation of saline solutions used with scleral rigid gas permeable contact lens wearers experiencing debris in the post lens tear reservoir

DETAILED DESCRIPTION:
One-month, approximately 36 subjects enrolled (~12/site), randomized, double-masked crossover trial.

Existing scleral rigid gas permeable (RGP) contact lens wearing subjects are randomly assigned (block) to different arms of the trial and receive different saline solutions for use sequentially for 2-week periods. The subjects will continue to wear their existing scleral GP lenses if lens fit is acceptable following an initial evaluation. Subjects will agree to complete a survey administered daily (via email) that will address contact lens wear time and subjective symptoms.

ELIGIBILITY:
Inclusion Criteria:•

* Daily wear large diameter (scleral) rigid gas permeable contact lens wearers in design with acceptable fit
* 18 years old or above.
* Agree to and sign Informed Consent.
* Correctable to at least 20/40 distance visual acuity in each eye.
* Presence of debris or "fogging" in post lens tear film reservoir (PLTR).

Exclusion Criteria:

* Extended wear contact lens wearers
* Require concurrent ocular medication.
* Grade 2 or more slit lamp findings (does not include fogging assessment).
* Eye injury or surgery within twelve weeks immediately prior to enrolment for this trial.
* Currently enrolled in an ophthalmic clinical trial.
* Pregnant or lactating
* Evidence of active ophthalmic disease or abnormality including glaucoma, chorioretinitis, central retinal artery or vein occlusion, intraocular or ocular infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Patient Subjective Symptoms and Wear Time Survey | 1 Month
  Participant Survey on Lens Comfort (based on a scale of 0 to 5), Symptoms (graded based on frequency (rarely/sometimes/often/always) and severity(slight/moderate/severe)), Total Wear Time (reported as hours per day) and How Many Times Lenses are Removed Daily (reported as number of times per day)

SECONDARY OUTCOMES:
Biomicroscopy Findings | 1 Month
  Edema, Bulbar Redness, Limbal Redness, Corneal Vascularization, Corneal Infiltrates, Palpebral Conjunctival Observations and Corneal Staining are evaluated on a grading scale of 0 to 4.
Visual Acuity | 1 Month
  Visual acuity (in units of Logmar) is evaluated with subject wearing habitual contact lenses.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Andre, MS, ABOe, Study Director — AVD Research
Locations (1):
- Andre Vision and Device Research, West Linn, Oregon, United States

IPD SHARING:
Plan to Share IPD: No